CLINICAL TRIAL: NCT00180115
Title: AML96 - Risk-Adapted and Randomized Postremission-Therapy for Adult Acute Myeloid Leukemia Patients. A Cooperative AML-Study of the German SHG-Study Group.
Brief Title: AML96 - Risk-Adapted and Randomized Postremission-Therapy for Adult Acute Myeloid Leukemia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MK1-191
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-07

CONDITIONS: Leukemia, Nonlymphoblastic, Acute
Keywords: acute myeloid leukemia; cytarabine postremission dosage; risk adapted treatment strategy; allogeneic stem cell transplantation; autologous stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

INTERVENTIONS:
Drug: Cytarabine Dosage

SUMMARY:
The AML96 study examines the feasibility of a risk-adapted postremission treatment strategy including related and unrelated allogeneic stem cell transplantation for high risk AML patients and related allogeneic and autologous stem cell transplantation for standard risk AML patients in a multi-center setting. Furthermore it randomizes patients between intermediate-dose Cytarabine vs high-dose Cytarabine within the first postremission-course.

DETAILED DESCRIPTION:
The AML96 study examines the feasibility of a risk-adapted postremission treatment strategy including related and unrelated allogeneic stem cell transplantation for high risk AML patients and related allogeneic and autologous stem cell transplantation for standard risk AML patients in a multi-center setting. Furthermore it randomizes patients between intermediate-dose Cytarabine vs high-dose Cytarabine within the first postremission-course.

ELIGIBILITY:
Inclusion Criteria:

* de novo or secondary acute myeloid leukemia of the FAB subtypes M0-M2 and M4-M7
* de novo or secondary myelodysplastic syndrome FAB subtypes RAEB and RAEB-T
* written informed consent

Exclusion Criteria:

* severe comorbidities
* severe uncontrolled complications of the leukemia
* previous therapy of leukemia/MDS
* HIV-Infection
* known relevant allergy against study medication
* pregnancy
* missing written informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1996-02; Study Completion 2008-11

PRIMARY OUTCOMES:
- rate of complete remission
- overall survival
- relapse-free survival

SECONDARY OUTCOMES:
- frequencies and grade of treatment side effects
- deaths within induction therapy
- deaths within postremission therapy
- feasibility according to dosages and time-intervals

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Ehninger, MD, Principal Investigator — University Hospital Carl Gustav Carus Dresden
Locations (1):
- Medical Department I, University Hospital Carl Gustav Carus, Dresden, Germany

REFERENCES:
- [Derived] Kunadt D, Stasik S, Metzeler KH, Rollig C, Schliemann C, Greif PA, Spiekermann K, Rothenberg-Thurley M, Krug U, Braess J, Kramer A, Hochhaus A, Scholl S, Hilgendorf I, Brummendorf TH, Jost E, Steffen B, Bug G, Einsele H, Gorlich D, Sauerland C, Schafer-Eckart K, Krause SW, Hanel M, Hanoun M, Kaufmann M, Wormann B, Kramer M, Sockel K, Egger-Heidrich K, Herold T, Ehninger G, Burchert A, Platzbecker U, Berdel WE, Muller-Tidow C, Hiddemann W, Serve H, Stelljes M, Baldus CD, Neubauer A, Schetelig J, Thiede C, Bornhauser M, Middeke JM, Stolzel F; A. M. L. Cooperative Group (AMLCG), Study Alliance Leukemia (SAL). Impact of IDH1 and IDH2 mutational subgroups in AML patients after allogeneic stem cell transplantation. J Hematol Oncol. 2022 Sep 5;15(1):126. doi: 10.1186/s13045-022-01339-8. PMID 36064577
- [Derived] Heidrich K, Thiede C, Schafer-Eckart K, Schmitz N, Aulitzky WE, Kramer A, Rosler W, Hanel M, Einsele H, Baldus CD, Trappe RU, Stolzel F, Middeke JM, Rollig C, Taube F, Kramer M, Serve H, Berdel WE, Ehninger G, Bornhauser M, Schetelig J; Study Alliance Leukemia (SAL). Allogeneic hematopoietic cell transplantation in intermediate risk acute myeloid leukemia negative for FLT3-ITD, NPM1- or biallelic CEBPA mutations. Ann Oncol. 2017 Nov 1;28(11):2793-2798. doi: 10.1093/annonc/mdx500. PMID 28945881
- [Derived] Herold T, Metzeler KH, Vosberg S, Hartmann L, Rollig C, Stolzel F, Schneider S, Hubmann M, Zellmeier E, Ksienzyk B, Jurinovic V, Pasalic Z, Kakadia PM, Dufour A, Graf A, Krebs S, Blum H, Sauerland MC, Buchner T, Berdel WE, Woermann BJ, Bornhauser M, Ehninger G, Mansmann U, Hiddemann W, Bohlander SK, Spiekermann K, Greif PA. Isolated trisomy 13 defines a homogeneous AML subgroup with high frequency of mutations in spliceosome genes and poor prognosis. Blood. 2014 Aug 21;124(8):1304-11. doi: 10.1182/blood-2013-12-540716. Epub 2014 Jun 12. PMID 24923295
- [Derived] Rollig C, Thiede C, Gramatzki M, Aulitzky W, Bodenstein H, Bornhauser M, Platzbecker U, Stuhlmann R, Schuler U, Soucek S, Kramer M, Mohr B, Oelschlaegel U, Stolzel F, von Bonin M, Wermke M, Wandt H, Ehninger G, Schaich M; Study Alliance Leukemia. A novel prognostic model in elderly patients with acute myeloid leukemia: results of 909 patients entered into the prospective AML96 trial. Blood. 2010 Aug 12;116(6):971-8. doi: 10.1182/blood-2010-01-267302. Epub 2010 May 4. PMID 20442365
- [Derived] Wandt H, Schakel U, Kroschinsky F, Prange-Krex G, Mohr B, Thiede C, Pascheberg U, Soucek S, Schaich M, Ehninger G. MLD according to the WHO classification in AML has no correlation with age and no independent prognostic relevance as analyzed in 1766 patients. Blood. 2008 Feb 15;111(4):1855-61. doi: 10.1182/blood-2007-08-101162. Epub 2007 Dec 4. PMID 18056840